CLINICAL TRIAL: NCT07197060
Title: Hypofractionated Radiotherapy With 3.5 Gy Per Fraction for Early Glottic Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Tarek mohamed, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: Hypofractionated 3.5 Gy Gc
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Early Glottic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Histologically confirmed squamous cell carcinoma of the glottis

SUMMARY:
Early-stage glottic carcinoma (T1-T2N0M0) is typically managed with either transoral laser microsurgery or definitive radiotherapy, both providing excellent local control rates and voice preservation outcomes. Radiotherapy remains a widely adopted non-invasive option, particularly for patients with bilateral disease or poor surgical candidacy. Traditionally, conventional fractionation schemes of 2.0-2.25 Gy per fraction over 6-7 weeks have been standard; however, emerging evidence supports the use of hypofractionated radiotherapy (HFRT) as an effective and more convenient alternative in this setting.

The unique anatomical confinement of early glottic tumors, along with their low propensity for lymphatic spread, makes them ideal candidates for dose escalation using hypofractionation. Several retrospective and prospective studies have demonstrated that higher doses per fraction (2.5-3.5 Gy) can yield comparable or superior local control rates compared to conventional regimens, without significantly increasing toxicity. The incorporation of modern techniques such as Intensity Modulated RadioTherapy (IMRT) and Simultaneous Integrated Boost (SIB) has further.enabled safe and precise delivery of escalated doses to the primary lesion while sparing nearby organs-at-risk (OARs)

Recent data have shown that a 3.5 Gy per fraction regimen (totaling 59.5 Gy in 17 fractions) achieves excellent tumor control with favorable toxicity profiles in selected patients. Additionally, omission of the posterior commissure from the elective target volume in the absence of direct tumor extension has been associated with reduced mucosal toxicity and improved patient-reported outcomes. Therefore,hypofractionated RT using 3.5 Gy per fraction offers a promising voice-preserving strategy in the treatment of early glottic cancer

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed squamous cell carcinoma of the glottis

  * Stage T1-T2N0M0 (AJCC 8th edition)
  * (based on clinical exam and imaging)
  * Age ≥ 18 years
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2
  * No prior radiotherapy or surgery to the larynx (except biopsy)
  * Adequate organ function and a life expectancy of at least 6 months
  * Ability to comply with follow-up schedule and complete voice assessments
  * Signed informed consent

Exclusion Criteria:

* • Prior head and neck irradiation

  * Nodal involvement or distant metastasis
  * Poor vocal cord mobility or subglottic extension
  * Severe comorbidities or life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with histologically confirmed squamous cell carcinoma of the glottisStage T1-T2N0M0 (AJCC 8th edition)based on clinical exam and imaging
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
local control rate | 2-year
  local control rate